CLINICAL TRIAL: NCT04042558
Title: A Multicentre Phase II, Open-label, Non-randomized Study Evaluating Platinum-Pemetrexed-Atezolizumab (+/- Bevacizumab) for Patients With Stage IIIB/IV Non-squamous Non-small Cell Lung Cancer With EGFR Mutations, ALK Rearrangement or ROS1 Fusion Progressing After Targeted Therapies
Brief Title: A Study Evaluating Platinum-Pemetrexed-Atezolizumab (+/-Bevacizumab) for Patients With Stage IIIB/IV Non-squamous Non-small Cell Lung Cancer With EGFR Mutations, ALK Rearrangement or ROS1 Fusion Progressing After Targeted Therapies
Acronym: GFPC 06-2018
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: GFPC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFPC 06-2018
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IV; EGFR Gene Mutation; ALK Gene Rearrangement Positive; ROS1 Gene Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Open-label, multicentre, non-randomized two parallel cohorts phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort with Bevacizumab (Experimental): 4 cycles of induction every 3 weeks with :
  * Carboplatin area under curve 6 mg/mL per minute per IV route or Cisplatin 75 mg/m² per IV route
  * Pemetrexed 500 mg/m² per IV route
  * Atezolizumab 1200 mg per IV route
  * Bevacizumab 15 mg/kg per IV route For patients without disease progression, treatment will be followed by maintenance therapy by Atezolizumab + Pemetrexed and Bevacizumab administered at the same dosage on 3-week cycles
  Interventions: Drug: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab
- Cohort without Bevacizumab (Experimental): 4 cycles of induction every 3 weeks with :
  * Carboplatin area under curve 6 mg/mL per minute per IV route or Cisplatin 75 mg/m² per IV route
  * Pemetrexed 500 mg/m² per IV route
  * Atezolizumab 1200 mg per IV route For patients without disease progression, treatment will be followed by maintenance therapy by Atezolizumab + Pemetrexed administered at the same dosage on 3-week cycles
  Interventions: Drug: Carboplatin + Pemetrexed + Atezolizumab

INTERVENTIONS:
Drug: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab — 4 cycles of induction every 3 weeks of cisplatine,pemetrexed, atezolizumab + bevacizumab and patients without disease progression, treatment will be followed by maintenance therapy by Atezolizumab + Pemetrexed +/- Bevacizumab administered at the same dosage on 3-week cycles
  Arms: Cohort with Bevacizumab
Drug: Carboplatin + Pemetrexed + Atezolizumab — Carboplatin + Pemetrexed + Atezolizumab
  Arms: Cohort without Bevacizumab

SUMMARY:
The objective of this study is to assess the efficacy of the combination of Platinum (carboplatin or cisplatin), Pemetrexed, Atezolizumab+/- Bevacizumab if eligible, in stage IIIB/IV non-squamous non-small cell lung cancer patients with progression-enhancing mutations following targeted therapies.

DETAILED DESCRIPTION:
In patients with an EGFR mutation, several phase III studies comparing EGFR tyrosine kinase inhibitors (TKIs) with chemotherapy have shown a benefit of TKI over chemotherapy, with no demonstrated benefit on overall survival. After a first line of treatment with a TKI, most patients progress and are eligible according to the mechanism of progression to a TKI of 3rd generation in case of T790M resistance or chemotherapy. In patients with ALK translocation, crizotinib has been shown to be beneficial in first line compared to a platinum doublet.Despite these major advances, most patients are progressing after targeted treatments and chemotherapy and are facing the problem of anti-PD1 / PDL1 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Subject affiliated to an appropriate social security system
* Signed informed consent before any trial related activities and according to local guidelines
* ECOG performance status of 0 or 1
* Histologically or cytologically confirmed, stage IIIB/IV non-squamous NSCLC (per the Union Internationale contre le Cancer/American Joint Committee on Cancer staging system, 7th edition).
* Patient with a sensitizing mutation in the EGFR gene must have experienced disease progression (during or after treatment) or intolerance to treatment with one or more EGFR TKIs, such as erlotinib, gefitinib, osimertinib or another EGFR TKI appropriate for the treatment of EGFR-mutant NSCLC. Patients with stage IIIB had to be not operable (that means not eligible for radiochemotherapy followed by a maintenance treatment by Durvalumab)
* Patient with an ALK fusion oncogene (confirmed in local laboratory) must have experienced disease progression (during or after treatment) or intolerance to treatment with one or more ALK inhibitors (i.e., crizotinib, alectinib, ceritinib) appropriate for the treatment of NSCLC in patients having an ALK fusion oncogene
* Patient with a ROS1 fusion oncogene (confirmed in local laboratory) must have experienced disease progression (during or after treatment) or intolerance to treatment with one or more ROS inhibitors (i.e., crizotinib,) appropriate for the treatment of NSCLC in patients having an ROS1 fusion oncogene
* No prior chemotherapy treatment for Stage IV non-squamous NSCLC except if less than 3 cycles, with treatment free-interval of at least 1 year from C1 since last chemotherapy
* Patient who has received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from C1since the last chemotherapy, radiotherapy, or chemoradiotherapy
* Patient with an history of asymptomatic CNS metastases is eligible, provided he meets all of the following criteria:

  * Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla, or spinal cord)
  * No ongoing requirement for corticosteroids as therapy for CNS disease
  * No stereotactic radiation within 7 days or whole-brain radiation within 14 days prior to inclusion
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function, defined by the following laboratory
* Adequate method of contraception during the treatment period and at least 5 months after the last dose of atezolizumab or 6 months after the last dose of chemotherapy

Exclusion Criteria:

Cancer-specific exclusions

* Active CNS metastases as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > or = 2 weeks prior to C1
* Leptomeningeal disease (Presence of cancer cells in cerebral CSF or MRI with leptomeningeal lesion strongly suspected of leptomeningeal disease )
* Uncontrolled tumour-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently); Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium > ULN)
* Malignancies other than NSCLC within 5 years prior to C1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)

General medical exclusions

* Women who are pregnant, lactating, or intending to become pregnant during the study
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are eligible for this study.
  * Patients with controlled Type 1 diabetes mellitus on a stable dose of insulin regimen are eligible for this study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are permitted provided that they meet the following conditions:
  * Rash must cover less than 10 percent of body surface area (BSA).
  * No acute exacerbations of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high-potency or oral steroids)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan; History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive test for HIV. All patients will be tested for HIV prior to C1 into the study; patients who test positive for HIV will be excluded from the study.
* Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
* Active tuberculosis
* Severe infections within 4 weeks prior to C1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Received therapeutic oral or IV antibiotics within 1 week prior to C1; Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to inclusion, unstable arrhythmias, or unstable angina
* Major surgical procedure other than for diagnosis within 28 days prior to C1 or anticipation of need for a major surgical procedure during the course of the study
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications
* Symptomatic brain metastases;
* Patients with illnesses or conditions that interfere with their capacity to understand, follow and/or comply with study procedures
* Concurrent participation in any therapeutic clinical trial
* Patient deprived of liberty or placed under the authority of a tutor
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Exclusion criteria related to medications

* Any approved anti-cancer therapy, including hormonal therapy within 7 days prior to C1 of study treatment.
* Treatment with any other investigational agent with therapeutic intent within 28 days prior to C1
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies

  * Patients who have had prior anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) treatment may be enrolled, provided the following requirements are met:
  * Last dose of anti-CTLA-4 at least 6 weeks prior to C1
  * No history of severe immune-related adverse effects from anti-CTLA-4 (NCI CTCAE Grade 3/4)
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferons, interleukin 2) within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to C1 ; Prior treatment with cancer vaccines is allowed.
* Treatment with systemic immunosuppressive medications (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to C1

Exclusion criteria related to chemotherapy

* History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds
* Patients with hearing impairment (cisplatin)
* Grade > or = 2 peripheral neuropathy as defined by NCI CTCAE v5.0 (cisplatin)
* CRCL < 60 mL/min for cisplatin or < 45 mL/min for carboplatin using the Cockcroft-Gault Method

Exclusion criteria related to Bevacizumab

* Medically uncontrolled hypertension (defined as PAS>150 and/or PAD >100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Clinically significant cardiovascular disease (within 6 months prior to C1) that is uncontrolled by medication or may interfere with administration of trial treatment:

  * Aortic aneurysm requiring surgical repair
  * Recent arterial thrombosis
  * Haemoptysis (>one-half teaspoon of bright red blood per episode (within one months prior to C1) (grade 2 haemoptysis)
* History of documented haemorrhagic diathesis or coagulopathy
* History of abdominal or tracheosphageal fistula or perforation within 6 months prior to C1
* Core biopsy or other minor surgical procedure within 7 days before bevacizumab
* Clinical signs or gastrointestinal obstruction or requirement for routine parenteral hydration, nutrition or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Major surgery within 28 days before C1
* Serious, non-healing wound, active ulcer or untreated bone fracture
* Proteinuria >1g/24h urine collection
* All patient with >2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate < or = 1g of protein in 24 hours.
* Known sensitivity to any component of bevacizumab
* Radiation therapy within 21 days before C1 (except Symptomatic lesions amenable to palliative radiotherapy)
* Adequate hematologic, liver, and renal function required (including creatinine clearance 45 mL/min at baseline and 45 mL/min before the start of any subsequent cycle using the Cockcroft-Gault Method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) according to RECIST 1.1 | After the end of 4 cycles (15 weeks)

SECONDARY OUTCOMES:
The progression-free survival (PFS) | 1 year
The overall survival | 1 year
The duration of response | 1 year

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU, Angers
  - Centre Hospitalier, Annecy
  - CHU-Hôpital MORVAN, Brest
  - CHU Lyon Louis Pradel, Bron
  - Centre François Baclesse, Caen
  - CHU Gabriel MONTPIED, Clermont-Ferrand
  - CHIC, Créteil
  - CHU, Grenoble
  - CHU Réunion St Denis, La Réunion
  - CHU Réunion St Pierre, La Réunion
  - CHD Vendée La Roche sur Yon, La Roche-sur-Yon
  - CHU, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CHU Lyon, Croix-Rousse,, Lyon
  - Hôpital Nord, Marseille
  - CHR Orléans, Orléans
  - Hopital Foch, Paris
  - institut Curie, Paris
  - HIA Percy, Percy
  - Hôpital Haut Lévêque,Centre François Magendie, Pessac
  - CHU, Pierre-Bénite
  - CHU, Rennes
  - CHU, Rouen
  - ICLN, St Priez en Jarez, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - HIA St Anne, Toulon
  - CHU, Toulouse
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre Hospitalier, Villefranche
  - HIA R.Picqué, Villenave-d'Ornon

REFERENCES:
- [Derived] Bylicki O, Tomasini P, Radj G, Guisier F, Monnet I, Ricordel C, Bigay-Game L, Geier M, Chouaid C, Daniel C, Swalduz A, Toffart AC, Doubre H, Peloni JM, Moreau D, Subtil F, Grellard JM, Castera M, Clarisse B, Martins-Lavinas PH, Decroisette C, Greillier L; GFPC. Atezolizumab with or without bevacizumab and platinum-pemetrexed in patients with stage IIIB/IV non-squamous non-small cell lung cancer with EGFR mutation, ALK rearrangement or ROS1 fusion progressing after targeted therapies: A multicentre phase II open-label non-randomised study GFPC 06-2018. Eur J Cancer. 2023 Apr;183:38-48. doi: 10.1016/j.ejca.2023.01.014. Epub 2023 Jan 31. PMID 36801605